CLINICAL TRIAL: NCT06139952
Title: Assessment of the Effect of Atorvastatin and N-acetyl Cysteine on Prevention of Contrast Induced Nephropathy in Patients Undergoing Coronary Angiography CIN
Brief Title: Ameliorating Contrast Induced Nephropathy After Coronary Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Sabry Hashem, Clinical Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease; Nephropathy; Toxic, Drugs
Keywords: Contrast Induced Nephropathy; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Kidney Diseases | interventions — Atorvastatin; Acetylcysteine; Saline Solution

STUDY DESIGN:
Intervention Model Description: A prospective single blinded multi armed randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-dose Atorvastatin group (Experimental): 40 patients will receive 80 mg Atorvastatin before coronary angiography and will receive adequate hydration using (1ml/kg/hr)
  Interventions: Drug: Atorvastatin 80mg
- N-acetyl cysteine group (Experimental): 40 patients will receive 200mg 3 times daily 2 days before coronary angiography and 2 days after and will receive adequate hydration using (1ml/kg/hr)
  Interventions: Drug: N-acetyl cysteine
- Control group (Active Comparator): 40 patients will receive adequate hydration using (1ml/kg/hr)
  Interventions: Drug: Atorvastatin 80mg; Drug: N-acetyl cysteine; Other: Normal Saline

INTERVENTIONS:
Drug: Atorvastatin 80mg — Atorvastatin 80mg taken Once before coronary angiography
  Arms: Control group; High-dose Atorvastatin group
Drug: N-acetyl cysteine — 200mg 3 times daily 2 days before coronary angiography
  Arms: Control group; N-acetyl cysteine group
Other: Normal Saline — adequate hydration using Normal Saline (1ml/kg/hr)
  Arms: Control group

SUMMARY:
Given the limited understanding of the impact of statin and N-acetyl cysteine use before angiography in preventing contrast-induced nephropathy (CIN), the objective of this study is to evaluate the effectiveness of atorvastatin in preventing CIN among patients undergoing coronary angiography.

DETAILED DESCRIPTION:
A multi armed randomized controlled clinical trial to be conducted from June 2023.According to inclusion and exclusion criteria, All patients presenting to the Cardiology department at Ain Shams University hospitals, will be assessed for eligibility. At least 120 patients subjected to elective CT coronary angiography who are at risk of developing contrast-induced renal failure will be enrolled. The participants will be assigned to Three groups (40 patients for each group):

* Three groups
* High-dose Atorvastatin group: 40 patients will receive 80 mg Atorvastatin before coronary angiography and will receive adequate hydration using (1ml/kg/hr)
* N-acetyl cysteine group: 40 patients will receive 200mg 3 times daily 2 days before coronary angiography and 2 days after and will receive adequate hydration using (1ml/kg/hr)
* Control group: 40 patients will receive adequate hydration using (1ml/kg/hr) The blood sample will be collected from all patients before the administration of contrast media and after 24 hours for assessment of the needed parameters.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective Coronary angiography who will receive coronary angiography contrast media.
* Must have at least two consecutive serum creatinine measurements (Before and after Contrast exposure)

Exclusion Criteria:

* Pregnant or lactating women
* Patients with Serum creatinine conc of >2.1 mg/Dl
* Patients undergoing emergency primary percutaneous coronary intervention for ST-segment elevation myocardial infarction.
* Prior exposure to contrast media within 7 days
* Contraindication for a high-dose statin, N-acetyl Cysteine prescription

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Contrast induced nephropathy (CIN) incidence | 24-48 hours after PCI
  Contrast-induced nephropathy was defined as an absolute increase of 0.5 mg/dL or a relative increase of >25% in creatinine levels 24-48 hours after the procedure.
  Contrast-induced nephropathy was defined as an absolute increase of 0.5 mg/dL or a relative increase of >25% in creatinine levels 24-48 hours after the procedure.
  Contrast-induced nephropathy was defined as an absolute increase of 0.5 mg/dL or a relative increase of >25% in creatinine levels 24-48 hours after the procedure.
  Contrast-induced nephropathy was defined as an absolute increase of 0.5 mg/dL or a relative increase of >25% in creatinine levels 24-48 hours after the procedure.
  Contrast-induced nephropathy was defined as an absolute increase of 0.5 mg/dL or a relative increase of >25% in creatinine levels

SECONDARY OUTCOMES:
Serum Creatinine (S.Cr) level | 48 hours after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- The Cardiovascular Hospital, Heliopolis, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang Y, Song M, Liu Y, Liu H, Sun L, Peng Y, Liu F, Venkatachalam MA, Dong Z. Renoprotective approaches and strategies in acute kidney injury. Pharmacol Ther. 2016 Jul;163:58-73. doi: 10.1016/j.pharmthera.2016.03.015. Epub 2016 Apr 22. PMID 27108948
- [Background] van der Molen AJ, Reimer P, Dekkers IA, Bongartz G, Bellin MF, Bertolotto M, Clement O, Heinz-Peer G, Stacul F, Webb JAW, Thomsen HS. Post-contrast acute kidney injury. Part 2: risk stratification, role of hydration and other prophylactic measures, patients taking metformin and chronic dialysis patients : Recommendations for updated ESUR Contrast Medium Safety Committee guidelines. Eur Radiol. 2018 Jul;28(7):2856-2869. doi: 10.1007/s00330-017-5247-4. Epub 2018 Feb 7. PMID 29417249
- [Background] Chong E, Poh KK, Lu Q, Zhang JJ, Tan N, Hou XM, Ong HY, Azan A, Chen SL, Chen JY, Ali RM, Fang WY, Lau TW, Tan HC. Comparison of combination therapy of high-dose oral N-acetylcysteine and intravenous sodium bicarbonate hydration with individual therapies in the reduction of Contrast-induced Nephropathy during Cardiac Catheterisation and Percutaneous Coronary Intervention (CONTRAST): A multi-centre, randomised, controlled trial. Int J Cardiol. 2015 Dec 15;201:237-42. doi: 10.1016/j.ijcard.2015.07.108. Epub 2015 Aug 5. PMID 26301645
- [Background] Ma WQ, Zhao Y, Wang Y, Han XQ, Zhu Y, Liu NF. Comparative efficacy of pharmacological interventions for contrast-induced nephropathy prevention after coronary angiography: a network meta-analysis from randomized trials. Int Urol Nephrol. 2018 Jun;50(6):1085-1095. doi: 10.1007/s11255-018-1814-0. Epub 2018 Feb 5. PMID 29404930
- [Background] Xie W, Liang X, Lin Z, Liu M, Ling Z. Latest Clinical Evidence About Effect of Acetylcysteine on Preventing Contrast-Induced Nephropathy in Patients Undergoing Angiography: A Meta-Analysis. Angiology. 2021 Feb;72(2):105-121. doi: 10.1177/0003319720950162. Epub 2020 Aug 24. PMID 32830526